CLINICAL TRIAL: NCT05880056
Title: A Prospective, Multicenter, Open-label, Single-arm Interventional Study of Bisoprolol (Nerkardou - Nerhadou International) 5 and 10 mg Oral Dissolvable Film (ODF) Treatment in Egyptian Patients With Essential Hypertension
Brief Title: Study of Bisoprolol (Nerkardou - Nerhadou International) 5 and 10 mg Oral Dissolvable Film (ODF) Treatment in Egyptian Patients With Essential Hypertension
Acronym: BETTER
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Genuine Research Center, Egypt (Industry)
Collaborators: Nerhadou International for pharmaceutical & Nutraceutical, Egypt (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRC/NE-CV/EG/39/IV
Record Dates: First submitted 2023-05-07; First posted 2023-05-30 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Intervention Model Description: The subject will initially administer once daily 5 mg bisoprolol (Nerkardou) oral dissolvable film (ODF) for 2 weeks. After the assessment of the subject being a responder, study medication will be maintained till week 12. Response will be assessed for each patient every 2 weeks and dose-titration will be done based on the response and PI decision at any visit. Then, for responders, once daily 5 mg bisoprolol (Nerkardou) oral dissolvable film (ODF will be administered for the subsequent 2 weeks. For non-responders once daily 10 mg bisoprolol (Nerkardou) oral dissolvable film (ODF) will be administered for the subsequent 2 weeks. Non responders patients on 10 mg will be shifted to other alternatives according to their merit and those patients will be included to intention to treat.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- (Nerkardou 5 mg) & (Nerkardou 10 mg) (Experimental): One ODF of bisoprolol 5 mg (Nerkardou 5 mg) Dosage form description: Bisoprolol oral dissolved film ODF: equivalent to 5 mg of bisoprolol fumarate.
  One ODF of bisoprolol 10 mg (Nerkardou 10 mg) Dosage form description: Bisoprolol oral dissolved film ODF: equivalent to 10 mg of bisoprolol fumarate.
  Interventions: Drug: Nerkardou (5 mg) & (10 mg)

INTERVENTIONS:
Drug: Nerkardou (5 mg) & (10 mg) — Bisoprolol oral dissolved film ODF(5 mg): equivalent to 5 mg of bisoprolol fumarate Bisoprolol oral dissolved film ODF (10 mg): equivalent to 10 mg of bisoprolol fumarate.
  Other Names: Bisoprolol oral dissolved film ODF (5 mg) & (10 mg)

SUMMARY:
The trial is designed to assess the safety and investigation of the efficacy of a single oral dose of bisoprolol (Nerkardou - Nerhadou) oral dissolvable film (ODF) 5 & 10 mg, and patients' compliance in the treatment of essential hypertension. This is a Phase IV, open-label, single-arm, prospective trial where subjects will receive:

1. Bisoprolol (Nerkardou) at an initial dose of 5 (mg) milligrams once daily for 2 weeks.
2. If the blood pressure would be greater than or equal to 130/80 mmHg after 2 weeks, then the dose will be titrated to 10 mg once daily (non-responders). Dose-Titration will be done at any follow-up visit based on the response.
3. The total duration of study treatment will be 12 weeks ±2 days, and the total sample size of the study will be 406 participants.

DETAILED DESCRIPTION:
The trial is designed to assess the safety and investigation of the efficacy of a single oral dose of bisoprolol (Nerkardou - Nerhadou) oral dissolvable film (ODF) 5 & 10 mg & patients' compliance in the treatment of essential hypertension. This is a Phase IV, open-label, single-arm, prospective trial where subjects will receive:

The subject will initially administer once daily 5 mg bisoprolol (Nerkardou) oral dissolvable film (ODF) for 2 weeks. After the assessment of the subject being a responder, study medication will be maintained till week 12. Response will be assessed for each patient every 2 weeks and dose-titration will be done based on the response and PI decision at any visit. Then, for responders, once daily 5 mg bisoprolol (Nerkardou) oral dissolvable film (ODF will be administered for the subsequent 2 weeks. For non-responders once daily 10 mg bisoprolol (Nerkardou) oral dissolvable film (ODF) will be administered for the subsequent 2 weeks. For those who are still not responding to the higher dose will be shifted to other alternatives according to their merit and they will be included to intention to treat.

A responder is defined by BP response, which is represented in the form of a ≥20 mmHg decreases in sitting through SBP and a ≥10 mmHg decreases in sitting through DBP, or a sitting through SBP of <130 mmHg and a sitting through DBP of <80 mmHg.

The total duration of study treatment will be 12 week (±2days). (Flow chart of trail design Appendix III) and the total sample size of the study will be 406 participants.

The trial has a duration of approximately 14 weeks, including:

1. Screening (assessments to determine eligibility for entry into the trial, occurring within 14 days to day 1 before treatment initiation (week -2) to (week 0).
2. Treatment duration (5 mg or 10 mg bisoprolol (Nerkardou) based on the response) (duration of 12 weeks); from Day 1 (week 1) to the end of day 84 ±2days (week 12 ±2days)
3. Premature withdrawal/ Early Discontinuation

ELIGIBILITY:
Inclusion Criteria:

1. The participant is willing and able to give informed consent for participation in the trial.
2. Male or Female, aged ≥ 21 and < 65 years.
3. The subject with Body mass index (BMI) greater than or equal to 18.5 and below 30 kg/m2
4. Newly diagnosed hypertensive patients with grade 1 and 2 are defined according to the recent ESC/ESH guidelines as follows:

   * Grade 1 hypertension: SBP 140 to 159mmHg and/or DBP 90 to 99mmHg
   * Grade 2 hypertension: SBP 160 to 179mmHg and/or DBP 100 to 109mmHg at screening.
5. Non-responders to the 1ST line of therapy for hypertension other than beta blocker and can be safely switched to Bisoprolol (Nerkardou) according to PI decision.
6. Subject doesn't have other comorbidity according to the assessment of the medical history, electrocardiogram (ECG), echocardiogram vital signs, physical examination, and laboratory results.
7. Subject with heart rate (HR) ≥ 80 (BPM) at baseline.
8. Female subjects in childbearing period, and not on a reliable contraceptive method must adhere to the recommended contraceptive methods as detailed in Appendix I.
9. Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the trial.

Exclusion Criteria:

1. Grade III hypertension or malignant hypertension (Hypertensive crisis: Systolic over 180 and/or diastolic over 120).
2. Subjects who are not legible to discontinue current antihypertensives such as calcium channel blockers (CCB), ACE- inhibitors, or diuretics for reasons other than hypertension, or responders to current therapy.
3. Subjects with heart rates less than (<)80 beats at rest.
4. Subjects with renal impairment (serum creatinine > 2.0 milligram per deciliter [mg/dL])
5. Subjects with unrecovered pulmonary edema
6. Subjects with a history of cardiovascular surgeries.
7. Significant history of hypersensitivity to bisoprolol, amlodipine, other dihydropyridines, or any related products (including excipients of the formulations)
8. Presence of diabetes mellitus
9. History or presence of asthma
10. Presence of significant gastrointestinal, liver, kidney disease, surgery, or any other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs or known to potentiate or predispose to undesired effects.
11. Use of any enzyme-modifying drugs, including strong inhibitors of CYP enzymes (such as cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem, and human immunodeficiency virus [HIV] antivirals) and strong inducers of CYP enzymes (such as barbiturates, carbamazepine, glucocorticoids, phenytoin, rifampin, St. John's wort or other herbal medicine known with effect on CYP enzymes) within 28 days before Day 1 of this trial
12. Acute conditions which might alter renal function (e.g., dehydration, severe infection)
13. History of suicidal tendency, history of, or disposition to seizures, state of confusion, clinically relevant psychiatric diseases
14. Positive pregnancy test (only for females of child-bearing potential), or females breastfeeding a child.
15. Consumption of large quantities of methylxanthine-containing beverages (more than 600 mg caffeine/day: 1 cup (250 mL) of coffee contains approximately 100 mg of caffeine, 1 cup of black or green tea contains approximately 30 mg and 1 glass of cola contains approximately 20 mg caffeine)
16. A participant with a life expectancy of fewer than 6 months, or inappropriate for the medication as defined in the Product Information such as acute heart failure or decompensation of heart insufficiency, that requires a therapy with inotropic agents; cardiogenic shock; AV block grade II or III, sick sinus syndrome, sinoatrial heart block; symptomatic bradycardia; symptomatic hypotonia; severe asthma bronchiolus or severe chronic obstructive airways disease; advanced stages of peripheral arterial disease or Raynaud's Syndrome; untreated pheochromocytoma, metabolic acidosis.
17. Participants who have participated in another research trial involving an investigational product in the past 12 weeks.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
The frequency of the first dose hypotension | At day 1 (week 1) within 1-4 hours of the first administration of 5& 10 mg doses
  The frequency of occurrence of the first dose hypotension, which is defined as a fall in systolic blood pressure of 20 mm Hg or more, or to a systolic blood pressure of less than 100 mm Hg, with or without associated symptoms.

SECONDARY OUTCOMES:
Identifying Bradycardia manifestation Assess the safety of Nerkardou ODF. | At day 14±2 (week 2), day 28±2 (week 4), day 42± 2 (week 6), day 56±2 (week 8), day 70±2 (week 10), and day 84±2 (week 12)
  Identify the number of patients with bradycardia manifestation, which is defined as heart rate reduction < 60 (bpm) after drug administration
Assess the safety of Nerkardou ODF. | At day 14±2 (week 2), day 28±2 (week 4), day 42±2 (week 6), day 56±2 (week 8), day 70±2 (week 10), and day 84±2 (week 12)
  Number of reported AEs
Investigate the efficacy of (Nerkardou) in treating patients with hypertension | At day 14±2 (week 2), day 28±2 (week 4), day 42±2 (week 6), day 56±2 (week 8), day 70±2 (week 10), and day 84±2 (week 12)
  Measuring the response rate for a patient's BP response, which is defined as a ≥20mmHg decrease in sitting through SBP and a ≥10mmHg decrease in sitting through DBP， or a sitting through SBP of <130mmHg and a sitting through DBP of <80mmHg
Investigate the overall response of (Nerkardou) in treating patients with hypertension | At the end of day 84±2 (week 12)
  The change of systolic blood pressure from baseline will be measured. The change of diastolic blood pressure from baseline will be measured
Measuring Patients' compliance to this dosage form, especially being easy to carry and easy to use | At day 14±2 (week 2), day 28±2 (week 4), day 42±2 (week 6), day 56±2 (week 8), day 70±2 (week 10), and day 84±2 (week 12)
  Doses returned will be counted at each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Bassem El-Zarif, MD, Ph.D, Principal Investigator — National Heart Institute, Cairo, Egypt; Khaled AlKhashab, MD, Ph.D, Principal Investigator — Faculty of Medicine, Fayoum University Hospital, Egypt; Heba Hamdy, MD, Ph.D, Principal Investigator — Faculty of Medicine, Beni-Suef University Hospital, Egypt
Locations (1):
- Al-Fayoum University Hospital, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fuchs FD, Whelton PK. High Blood Pressure and Cardiovascular Disease. Hypertension. 2020 Feb;75(2):285-292. doi: 10.1161/HYPERTENSIONAHA.119.14240. Epub 2019 Dec 23. PMID 31865786
- [Background] NCD Risk Factor Collaboration (NCD-RisC). Worldwide trends in hypertension prevalence and progress in treatment and control from 1990 to 2019: a pooled analysis of 1201 population-representative studies with 104 million participants. Lancet. 2021 Sep 11;398(10304):957-980. doi: 10.1016/S0140-6736(21)01330-1. Epub 2021 Aug 24. PMID 34450083
- [Background] Channaraya V, Marya RK, Somasundaram M, Mitra D, Tibrewala KD; BRIGHT investigators. Efficacy and tolerability of a beta-1 selective beta blocker, bisoprolol, as a first-line antihypertensive in Indian patients diagnosed with essential hypertension (BRIGHT): an open-label, multicentric observational study. BMJ Open. 2012 May 14;2(3):e000683. doi: 10.1136/bmjopen-2011-000683. Print 2012. PMID 22586283
- [Background] Hostalek-Gottwald U, Gaciong Z. A growing evidence base for the fixed-dose combination of bisoprolol and amlodipine to manage hypertension. Curr Med Res Opin. 2022 Jul;38(7):1047-1053. doi: 10.1080/03007995.2022.2072087. Epub 2022 May 13. PMID 35510372
- [Background] Mancia G, Laurent S, Agabiti-Rosei E, Ambrosioni E, Burnier M, Caulfield MJ, Cifkova R, Clement D, Coca A, Dominiczak A, Erdine S, Fagard R, Farsang C, Grassi G, Haller H, Heagerty A, Kjeldsen SE, Kiowski W, Mallion JM, Manolis A, Narkiewicz K, Nilsson P, Olsen MH, Rahn KH, Redon J, Rodicio J, Ruilope L, Schmieder RE, Struijker-Boudier HA, Van Zwieten PA, Viigimaa M, Zanchetti A. Reappraisal of European guidelines on hypertension management: a European Society of Hypertension Task Force document. Blood Press. 2009;18(6):308-47. doi: 10.3109/08037050903450468. No abstract available. PMID 20001654
- [Background] Mancia G, Kreutz R, Brunstrom M, Burnier M, Grassi G, Januszewicz A, Muiesan ML, Tsioufis K, Agabiti-Rosei E, Algharably EAE, Azizi M, Benetos A, Borghi C, Hitij JB, Cifkova R, Coca A, Cornelissen V, Cruickshank JK, Cunha PG, Danser AHJ, Pinho RM, Delles C, Dominiczak AF, Dorobantu M, Doumas M, Fernandez-Alfonso MS, Halimi JM, Jarai Z, Jelakovic B, Jordan J, Kuznetsova T, Laurent S, Lovic D, Lurbe E, Mahfoud F, Manolis A, Miglinas M, Narkiewicz K, Niiranen T, Palatini P, Parati G, Pathak A, Persu A, Polonia J, Redon J, Sarafidis P, Schmieder R, Spronck B, Stabouli S, Stergiou G, Taddei S, Thomopoulos C, Tomaszewski M, Van de Borne P, Wanner C, Weber T, Williams B, Zhang ZY, Kjeldsen SE. 2023 ESH Guidelines for the management of arterial hypertension The Task Force for the management of arterial hypertension of the European Society of Hypertension: Endorsed by the International Society of Hypertension (ISH) and the European Renal Association (ERA). J Hypertens. 2023 Dec 1;41(12):1874-2071. doi: 10.1097/HJH.0000000000003480. Epub 2023 Sep 26. PMID 37345492
- [Background] Deedwania P. Hypertension, dyslipidemia, and insulin resistance in patients with diabetes mellitus or the cardiometabolic syndrome: benefits of vasodilating beta-blockers. J Clin Hypertens (Greenwich). 2011 Jan;13(1):52-9. doi: 10.1111/j.1751-7176.2010.00386.x. Epub 2010 Nov 8. PMID 21214722
- [Background] Prichard BN, Cruickshank JM, Graham BR. Beta-adrenergic blocking drugs in the treatment of hypertension. Blood Press. 2001;10(5-6):366-86. doi: 10.1080/080370501753400665. PMID 11822540
- [Background] Dutta A, Lanc R, Begg E, Robson R, Sia L, Dukart G, Desjardins R, Yacobi A. Dose proportionality of bisoprolol enantiomers in humans after oral administration of the racemate. J Clin Pharmacol. 1994 Aug;34(8):829-36. doi: 10.1002/j.1552-4604.1994.tb02047.x. PMID 7962671
- [Background] Minushkina LO. [Bisoprolol: opportunities in the treatment of hypertension]. Kardiologiia. 2012;52(6):80-5. Russian. PMID 22839675
- [Background] Wee Y, Burns K, Bett N. Medical management of chronic stable angina. Aust Prescr. 2015 Aug;38(4):131-6. doi: 10.18773/austprescr.2015.042. Epub 2015 Aug 3. PMID 26648642
- [Background] Johns TE, Lopez LM. Bisoprolol: is this just another beta-blocker for hypertension or angina? Ann Pharmacother. 1995 Apr;29(4):403-14. doi: 10.1177/106002809502900412. PMID 7633020
- [Background] Lancaster SG, Sorkin EM. Bisoprolol. A preliminary review of its pharmacodynamic and pharmacokinetic properties, and therapeutic efficacy in hypertension and angina pectoris. Drugs. 1988 Sep;36(3):256-85. doi: 10.2165/00003495-198836030-00002. PMID 2903820
- [Background] Tjandrawinata RR, Setiawati E, Yunaidi DA, Santoso ID, Setiawati A, Susanto LW. Bioequivalence study of two formulations of bisoprolol fumarate film-coated tablets in healthy subjects. Drug Des Devel Ther. 2012;6:311-6. doi: 10.2147/DDDT.S36567. Epub 2012 Oct 30. PMID 23139624
- [Background] Baxter AJ, Spensley A, Hildreth A, Karimova G, O'Connell JE, Gray CS. Beta blockers in older persons with heart failure: tolerability and impact on quality of life. Heart. 2002 Dec;88(6):611-4. doi: 10.1136/heart.88.6.611. PMID 12433890
- [Background] Davidov ME, Singh SP, Vlachakis ND, Blumenthal JB, Simon JS, Bryzinski BS, Koury KJ, Alemayehu D. Bisoprolol, a once-a-day beta-blocking agent for patients with mild to moderate hypertension. Clin Cardiol. 1994 May;17(5):263-8. doi: 10.1002/clc.4960170509. PMID 8004841
- See also: Hypertension [Internet]. World Health Organization. 2023 [cited 2023 Dec 13]. — http://www.who.int/news-room/fact-sheets/detail/hypertension
- See also: Raised cholesterol [Internet]. World Health Organization. [cited 2023 Dec 13] — http://www.who.int/data/gho/indicator-metadata-registry/imr-details/3236
- See also: World Health Organization. Egypt STEPS Survey 2017. 2017 — http://cdn.who.int/media/docs/default-source/ncds/ncd-surveillance/data-reporting/egpyt/steps/egypt-steps-survey-2017-facts-and-figures.pdf?sfvrsn=f4dd4788_2&download=true
- See also: Bisoprolol Pharmacokinetics — http://www.ncbi.nlm.nih.gov/books/NBK551623/?report=reader